CLINICAL TRIAL: NCT05565898
Title: Diagnostic Performance of PET/CT Vs Bone Marrow Biopsy in Exclusion of BM Infiltration for Initial Staging of Lymphoma
Brief Title: PET/CT Vs Bone Marrow Biopsy in Exclusion of Bone Marrow Infiltration for Initial Staging of Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Sharef Eid Ahmed, Principle investigator, Assiut University
Other Study IDs: PET/CT In lymphoma
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma
Keywords: lymphoma; PET/CT; Bone Marrow
MeSH Terms: conditions — Lymphoma | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow biopsy pathology
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: positron emission tomography for exclusion of bone marrow infiltration in lymphoma — compare the diagnostic accuracy of PET/CT scan against Bone Marrow Biopsy in detection of bone marrow involvement for staging of lymphoma

SUMMARY:
lymphoma is a common malignancy in the developed world. the two main categories of lymphoma are non-Hodgkin lymphoma and non-Hodgkin lymphoma. Bone marrow biopsy (BMB) is the most direct method of detecting lymphoma infiltration, however it is an invasive procedure. 18 fluro-2deoxy-D glucose PET/CT is a non-invasive examination that can comperhensively evaluate the state of bone marrow (BM) with extremely high sensitivity in detecting bone marrow infiltration of lymphoma.

DETAILED DESCRIPTION:
Lymphoma is a common malignancy in the developed world. Many subtypes of lymphomas are known. The two main categories of lymphoma are the non-Hodgkin lymphoma (NHL) (90% of cases) and Hodgkin lymphoma (HL) (10%). Lymphoma makes up 3-4% of all cancers, making them as a group the seventh-most common form.

Bone marrow biopsy is the most direct method of detecting lymphoma infiltration, however, it is an invasive procedure which is accompanied by several complications such as pain, hemorrhage and may miss marrow involvement if infiltration is patchy, or not taken from a part of the marrow that is involved.

18fluoro-2-deoxy-D-glucose (FDG) positron emission tomography/computed tomography (PET/CT) is a non-invasive examination that can comprehensively evaluate the state of bone marrow with extremely high sensitivity in detecting bone marrow infiltration of lymphoma and can replace bone marrow biopsy.

At this moment, there is no clear international guideline between the indications of PET-CT and bone marrow biopsy, but there is interest in using the PET/CT findings to either supplement or even replace the BMB in the evaluation of BM involvement in lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Initial diagnosed patient not receiving treatment.
* Baseline bone marrow biopsy.
* Baseline PET/CT.
* The period between performing PET/CT and bone marrow biopsy is maximum 30 days and without lymphoma treatment between the studies.

Exclusion Criteria:

* Patient receiving chemotherapy or corticosteroid before doing PET/CT and BMB.
* patients with known concomitant malignancy.
* patients who received hemopoietic growth factor injections less than 48 hours before the PET/CT.
* patients with previously known and treated lymphoma.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient Intially diagnosed with lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Comparison between PET/CT and BMB in detection of bone marrow involvement | 30 days between initial bone marrow biopsy and initial PET/CT before starting treatment for lymphoma
  Compare the diagnostic accuracy of PET/CT scan against Bone Marrow Biopsy in detection of bone marrow involvement for staging of lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Taha Z. Mohran, M.D, Study Chair — Assiut university- Faculty of Medicine-Department of Clinical Oncology and Nuclear Medicine; Nahla M Mahmoud, M.D, Study Director — Assiut university- Faculty of Medicine-Department of Clinical Oncology and Nuclear Medicine; Maha Kh Mahmoud, M.D, Study Director — Assiut university- Faculty of Medicine-Department of Clinical Oncology and Nuclear Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tang HJ. [PET/CT Image Values in Clinical Staging of the Patients with Non-Hodgkin's Lymphoma]. Zhongguo Shi Yan Xue Ye Xue Za Zhi. 2015 Aug;23(4):1030-3. doi: 10.7534/j.issn.1009-2137.2015.04.024. Chinese. PMID 26314440
- [Background] Angelopoulou MK, Mosa E, Pangalis GA, Rondogianni P, Chatziioannou S, Prassopoulos V, Moschogianni M, Tsirkinidis P, Asimakopoulos JV, Konstantinou I, Tsourouflis G, Sachanas S, Yiakoumis X, Boutsikas G, Arapaki M, Gainaru G, Kyrtsonis MC, Siakantaris MP, Datseris I, Panayiotidis P, Konstantopoulos K, Vassilakopoulos TP. The Significance of PET/CT in the Initial Staging of Hodgkin Lymphoma: Experience Outside Clinical Trials. Anticancer Res. 2017 Oct;37(10):5727-5736. doi: 10.21873/anticanres.12011. PMID 28982893
- [Background] Metser U, Dudebout J, Baetz T, Hodgson DC, Langer DL, MacCrostie P, Mak V, Tau N. [18 F]-FDG PET/CT in the staging and management of indolent lymphoma: A prospective multicenter PET registry study. Cancer. 2017 Aug 1;123(15):2860-2866. doi: 10.1002/cncr.30672. Epub 2017 Mar 13. PMID 28295218
- [Background] Berthet L, Cochet A, Kanoun S, Berriolo-Riedinger A, Humbert O, Toubeau M, Dygai-Cochet I, Legouge C, Casasnovas O, Brunotte F. In newly diagnosed diffuse large B-cell lymphoma, determination of bone marrow involvement with 18F-FDG PET/CT provides better diagnostic performance and prognostic stratification than does biopsy. J Nucl Med. 2013 Aug;54(8):1244-50. doi: 10.2967/jnumed.112.114710. Epub 2013 May 14. PMID 23674577
- [Background] Liden Y, Landgren O, Arner S, Sjolund KF, Johansson E. Procedure-related pain among adult patients with hematologic malignancies. Acta Anaesthesiol Scand. 2009 Mar;53(3):354-63. doi: 10.1111/j.1399-6576.2008.01874.x. PMID 19243321